CLINICAL TRIAL: NCT03318107
Title: Pilot Study of Ultrasound and Photoacoustic Imaging for Assessing Treatment Response of Cervical Cancer Patients
Brief Title: Ultrasound and Photoacoustic Imaging for Cervical Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201710024
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Cervical Cancer; Cancer of the Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transvaginal probe (Photoacoustic + ultrasound imaging) (Experimental): * A transvaginal imaging probe using ultrasound and photoacoustic imaging will be inserted into the vagina and will use different frequencies of lights to create images
  * This will occur before the first standard of care treatment, mid-treatment, end of treatment, and approximately 3 months after the end of treatment for a total of 4 imaging time points
  Interventions: Device: Transvaginal probe using photoacoustic and ultrasound imaging

INTERVENTIONS:
Device: Transvaginal probe using photoacoustic and ultrasound imaging — -Four optical wavelengths of 730nm, 780nm, 800 nm, and 830 nm will be used to acquire data

SUMMARY:
The investigators have developed co-registered transvaginal photoacoustic and ultrasound (US) imaging techniques that allow them to visualize ovarian tumor structure and functional changes simultaneously, which may potentially reveal early tumor angiogenesis development or residual tumors after systemic treatment that is not available by US alone. The ability to detect early angiogenesis changes, as well as tumor morphology changes using a non-invasive imaging modality will greatly enhance the care for patients. The investigators plan to explore these techniques in monitoring cervical cancer treatment response and conduct pilot feasibility studies.

ELIGIBILITY:
* Diagnosis of cervical cancer of any stage that will be treated with radiation therapy and concurrent chemotherapy.
* At least 18 years of age.
* Not pregnant and/or breastfeeding.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete the imaging protocol | Approximately 18 weeks

SECONDARY OUTCOMES:
Reduction rate of tumor angiogenesis | 3 months after completion of standard of care treatment (approximately 18 weeks)
  * The reduction rate of tumor angiogenesis of clinical responders and non-responders will be analyzed
  * Responders and non-responders will be determined by standard of care PET imaging based on F18-FDG uptake, 3 months after completion of treatment
Charge pattern of blood oxygen saturation | 3 months after completion of standard of care treatment (approximately 18 weeks)
  * The charge pattern of blood oxygen saturation of clinical responders and non-responders will be analyzed
  * Responders and non-responders will be determined by standard of care PET imaging based on F18-FDG uptake, 3 months after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Perry W Grigsby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu